CLINICAL TRIAL: NCT06961539
Title: The Effect on Pain, Anxiety and Sleep Levels of Virtual Visiting in the Cardiovascular Surgery Intensive Care Unit: A Randomized Controlled Trial
Brief Title: "The Effect of Virtual Visitation in the Intensive Care Unit on Pain, Anxiety, and Sleep Levels"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülay Karatay, Graduate Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBU-SBF-GK-01
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Pain; Cardiovascular surgery; Anxiety; virtual visiting; sleep
MeSH Terms: conditions — Coronary Artery Disease; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group with virtual visits (Experimental): In this group, in addition to face-to-face visits in the intensive care unit after cardiac surgery, virtual visits were conducted with the patients' relatives via WhatsApp (a type of smartphone app) through a smartphone by the applying researcher, totaling five minutes. These visits were conducted twice on the first day after surgery, at 10:00 AM (Ante Meridiem) and 10:00 PM ( Post Meridiem)."
  Interventions: Other: The group with virtual visits
- The group without virtual visits (No Intervention): In this group, patients received a face-to-face visit once a day at 1:00 PM (Post Meridiem) on the first day after surgery, according to the clinic's routine. The scales used in the study were applied at the same time interval as in the intervention group."

INTERVENTIONS:
Other: The group with virtual visits — On the first day after open-heart surgery in the intensive care unit, in addition to face-to-face visits, video calls were made through the researcher's phone in the morning and evening."
  Arms: The group with virtual visits

SUMMARY:
Patients in the intensive care unit after cardiovascular surgery face not only complications related to the surgical procedure but also emotional distress due to separation from their loved ones.

Because of infection control measures, visitor restrictions are enforced in intensive care units, which may further contribute to patient stress.

This study aims to evaluate the effect of scheduled virtual visitation in the intensive care environment on patients' postoperative pain, anxiety, and sleep levels.

DETAILED DESCRIPTION:
Cardiovascular diseases are a group of disorders of the heart and blood vessels, causing an estimated 17.9 million deaths globally each year, and are among the leading causes of death worldwide.Coronary artery bypass graft (CABG) surgery, considered a last-resort treatment option in terms of cardiovascular disease risk factors, is a costly intervention; however, it has shown an increasing trend in its application over the past 50 years and remains the most commonly performed cardiac surgical procedure worldwide.Postoperative complications not only negatively affect the patient's recovery process but also lead to an increase in healthcare costs (9). Common issues related to surgery and anesthesia include changes in the respiratory, circulatory, and neurological systems, as well as discomfort such as pain, nausea, and vomiting.Additionally, the isolated environment of the intensive care unit can lead to various emotional problems such as delirium, anxiety, depression, spiritual distress, pain, and sleep disturbances, alongside physiological complications.

Technology provides significant convenience in all aspects of our lives. The use of technological applications in healthcare is becoming increasingly widespread and is preferred by patients, their relatives, and healthcare professionals. Surgical procedures can lead to both physical and psychological complications in patients. The fact that the patient is in a foreign environment, such as an intensive care unit, and cannot see their loved ones at will, adds an extra source of stress for the patient.

Virtual visitation in the intensive care unit is not only an easy, cost-effective, and reliable method, but it can also have positive psychological effects for both the patient and their family. The virtual visitation application can be used as an alternative option for relatives who cannot visit the hospital due to distance, cost, illness, or other responsibilities, and as a result, cannot meet with their loved one. From the patient's perspective, being able to meet with a relative at any time during treatment in the foreign and complex environment of the intensive care unit has been shown to have positive effects in the studies in the literature. However, in the related literature review, it was observed that virtual visitation was only used during the COVID-19 (Coronavirus Disease 2019) pandemic, and there were no studies that combined virtual visits with face-to-face visits. Virtual visitation should also be an alternative visitation option for patients who undergo major surgeries, such as coronary artery bypass graft (CABG) surgery, and require postoperative follow-up in the intensive care unit. No studies have been found evaluating pain, anxiety, and sleep levels in CABG patients after virtual visits, and it is expected that this study will contribute to the literature in this regard.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 and above,
* Underwent elective coronary artery bypass graft surgery,
* Conscious, extubated, and hemodynamically stable,
* Glasgow Coma Scale score of 15,
* Followed in the intensive care unit for at least 48 hours after surgery,
* Patients who agreed to participate in the study.

Exclusion Criteria:

* Patients with psychiatric disorders and using medication,
* Illiterate patients,
* Patients without a relative who can conduct the virtual visit,
* Patients with communication problems.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
The Numeric Rating Scale | one day
  The Numerical Rating Scale is a unidimensional scale used to measure pain intensity, with numerical values ranging from 0 to 10. The patient is asked to choose the number that best reflects the pain intensity, where 0 = no pain and 10 = the worst (intolerable) pain."

SECONDARY OUTCOMES:
The State-Trait Anxiety Inventory" | one day
  The inventory consists of two subscales: State Anxiety and Trait Anxiety. The State Anxiety Inventory measures how an individual expresses themselves in the current situation, while the Trait Anxiety Inventory measures how the individual expresses themselves in general, not in a specific moment. The State Anxiety Inventory consists of a total of 20 items. Each item in the inventory uses a four-point Likert scale: "(1) not at all," "(2) a little," "(3) quite a bit," and "(4) completely," with reverse scoring applied to items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The total score obtained from the inventory ranges from 20 to 80. A higher score on the inventory indicates a higher level of anxiety in the individual.

OTHER OUTCOMES:
The Richard-Campbell Sleep Scale | two day
  The scale consists of six items that assess factors affecting sleep patterns, such as the depth of night sleep, sleep onset latency, frequency of awakenings, duration of wakefulness, sleep quality, and the noise level in the environment. The scale score ranges from "0-25," indicating "very poor sleep," to "76-100," indicating "very good sleep." The total score evaluation is based on five items, with the sixth item not included in the total score calculation. The higher the scale score, the more positive the improvement in the individual's sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Karatay, Principal Investigator — Saglik Bilimleri Universitesi; Elif Gezginci Akpınar, Assoc. Prof., Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Hamidiye Institute of Health Sciences, University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No